CLINICAL TRIAL: NCT04248309
Title: The Effect of Serum Progesterone Level on Day 3 in HRT-FET Cycles on the Clnical Outcome: a Randomized Controlled Study
Brief Title: Serum Progesterone Level in HRT-FET：a RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Haiyan Lin, Principal investigator, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-HRT-P-05
Record Dates: First submitted 2020-01-27; First posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Progesterone,Hormone Replacement Thawed Embryo Transfer Cycles

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A1 (Experimental): The included patient should test serum progesterone level on D3 no matter which day perform the embryo transfer. According to the progesterone level, there are two groups, Group A: serum progesterone <7.24ug/L, followed by randomized A1: plus additional treatment（intramuscular progesterone 20-40mg from D3 ）
  Interventions: Drug: intramuscular progesterone 20-40mg from D3 until pregnancy test
- A2 (No Intervention): The included patient should test serum progesterone level on D3 no matter which day perform the embryo transfer. According to the progesterone level, there are two groups, Group A: serum progesterone <7.24ug/L, followed by randomized A2：without additional treatment
- B (No Intervention): Group B：serum progesterone ≥7.24ug/L， without additional treatment

INTERVENTIONS:
Drug: intramuscular progesterone 20-40mg from D3 until pregnancy test — serum progesterone <7.24ug/L, followed by randomized A1: plus additional treatment（intramuscular progesterone 20-40mg from D3 ）
  Arms: A1

SUMMARY:
In the window of implantation, progesterone plays an important role. Sufficient serum progesterone is basic for ongoing pregnancy. Vaginal progesterone is more and more widely used in ART. As it has no hepatic first pass effect. What is the optimal serum level for pregnancy when use vaginal progesterone is not known yet? Hormone replacement therapy- FET is the optimal strategy to explore this question. There are some retrospective studies showed that the serum progesterone level on embryo transfer day (D3 or D5) or pregnancy test day (D14) lower than 10-11ng/ml is significantly associated with ongoing pregnancy rate in HRT-FET cycles. This prospective study is designed to compare the ongoing pregnancy rate between different serum progesterone levels on D3 and to explore the intervention of additional progesterone supplement since D3 is helpful in HRT-FET cycles.

ELIGIBILITY:
Inclusion Criteria:

1. HRT-FET cycles，including GnRHa-HRT-FET
2. Age<41 years old
3. BMI<30kg/m2
4. TSH and PRL normal
5. Endometrium thickness ≥8mm on D0 6） embryo transfer completed with at least 1 top-quality embryo (7-9 cell Grade 1 or D5 beyond grade 3 ) 7） Scandalized luteal phase support： transvaginal progesterone 0.2 tid with or without oral progesterone 10mg bid 8） included once for every patient

Exclusion Criteria:

1. history of Moderate and Severe uterine adhesion；
2. presence of hydrosapinx diameter >2cm
3. Endometrosis at stage III-IV
4. Recurrent implantation failure (>3 times of embryo transfer cycle)

Ages: 20 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 423 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 10 weeks after embryo transfer
  beyond pregnancy week 12 in HRT-FET cycles

SECONDARY OUTCOMES:
Clinical pregnancy rate | 10 weeks after embryo transfer
  intrauterine gestational sacs by ultrasound

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Haiyan L, Gang Y, Yu L, Lin L, Xiaoli C, Qingxue Z. Does serum progesterone level impact the ongoing pregnancy rate in frozen embryo transfer under artificial preparation with vaginal progesterone? Study protocol for a randomized controlled trial. Trials. 2022 Jan 3;23(1):3. doi: 10.1186/s13063-021-05953-8. PMID 34980220